CLINICAL TRIAL: NCT01171391
Title: An Open Label, Dose Escalation Study to Assess Intra-Subject Dose Response to VA106483 in Female Subjects
Brief Title: VA106483 Dose Response in Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vantia Ltd (Industry)
Responsible Party: Chief Medical Officer, Vantia Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 483-007
Record Dates: First submitted 2010-07-19; First posted 2010-07-28 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Nocturia
Keywords: Nocturia; Pharmacokinetics; Pharmacodynamics; Water-loading; Females
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- VA106483 1mg (Experimental)
  Interventions: Drug: VA106483
- VA106483 2mg (Experimental)
  Interventions: Drug: VA106483
- VA106483 4mg (Experimental)
  Interventions: Drug: VA106483
- Sugar pill (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VA106483 — 1 mg VA106483 on Day 3, 2 mg VA106483 on Day 5 and 4 mg VA106483 on Day 7
  Arms: VA106483 1mg; VA106483 2mg; VA106483 4mg
Other: Placebo — Placebo on Day 1
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to describe the pharmacokinetics and pharmacodynamics of VA106483 in female subjects.

DETAILED DESCRIPTION:
Nocturia, defined as waking to void at least once per night between periods of sleep, is a common complaint and shows an age-dependent increase in both prevalence and severity (number of nocturnal voids). The most common causes are detrusor over-activity, reduced nighttime functional bladder capacity, and nocturnal polyuria.

VA106483 is a selective vasopressin V2-receptor agonist in development for nocturia. VA106483 is a non-peptide drug that displays much improved oral availability over desmopressin and low dependence on glomerular filtration for its elimination.

VA106483 has been administered to 184 subjects (including healthy adult subjects [males and females], children [males and females] with nocturia and 48 elderly males [aged 65 years and over]). It has been administered as single doses both intravenously, up to doses of approximately 250 mg and orally up to 50 mg It is also being investigated in approximately 123 male subjects (two-thirds on active medication, one third on placebo) with nocturia in a current study with dosing for up to 8 weeks.

This intra-subject dose escalation study has previously been conducted in 10 elderly male subjects to determine whether subjects demonstrated a dose-dependent pharmacokinetic and pharmacodynamic (urine osmolality and diuresis) response and whether the dose of VA106483 could be titrated within an individual patient to achieve optimal clinical response in clinical practice. Given that to date, only 8 females have been exposed to VA106483, the purpose of this study is to confirm that the described duration of pharmacokinetics and pharmacodynamics of VA106483 in males is similar in females.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects 40 years and above
* BMI 18 to 32 kg/m2
* Using adequate contraception and providing negative pregnancy tests pre-dose
* In good health as determined by medical history and screening tests
* Subject is willing and able to abstain from alcohol and caffeine-containing food and beverages 72 hours prior to dosing and throughout the study
* Provide written, informed consent

Exclusion Criteria:

* Pregnancy or lactation
* Evidence of serious pathology or diseases including heart, hormone, liver and kidney, psychiatric and neurological problems, including syndrome of inappropriate antidiuretic hormone secretion, polydipsia or diabetes insipidus
* Likely to be hypersensitive to VA106483
* History of any relevant allergy
* Participation in a clinical study within 30 days
* Donation of blood (500 mL) within 60 days prior to dosing
* A history of alcohol abuse or drug addiction
* Positive results for HIV, HBV or HCV or drugs of abuse
* Currently taking any diuretics or clinically significant cytochrome 3A4 inhibitors or inducers
* Use of any non-prescription preparation within 72 hours prior to dosing, with the exception of ibuprofen, and acetaminophen used at recommended doses
* Treatment within the previous 3 months of drugs known to have a well defined potential for hepatoxicity
* Current smokers or recent ex-smokers
* Other protocol defined eligibility criteria may apply

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 10 days
  VA106483 plasma concentration pre-dose over a 24hr post-dose period to assess pharmacokinetics of each dose level

SECONDARY OUTCOMES:
Pharmacodynamics | 10 days
  Urine volume and osmolality
Safety and Tolerability | 10 days
  AEs, laboratory safety tests, vital signs and ECG, physical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Schutz, Principal Investigator — Quintiles Phase I Services
Locations (1):
- Quintiles Phase I Services, Overland Park, Kansas, United States